CLINICAL TRIAL: NCT05238935
Title: Do All Patients With Congenital Hip Dysplasia Corrected Operativell Need Physiotherapy
Brief Title: Do All Patients With Congenital Hip Dysplasia Corrected Operatively Need Physiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Dr. Hadeel Alsaleh, physiotherapy and rehabilitation specialist, Ministry of Health, Kuwait
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1920
Record Dates: First submitted 2022-01-19; First posted 2022-02-14 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Developmental Dysplasia of the Hip
Keywords: DDH; physiotherapy; rehabilitation; home program
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Intervention Model Description: Individuals who meet the inclusion criteria and had their guardian agreed to volunteer will be included in the study by signing the Informed Voluntary Consent Form and will be randomly allocated into either control group or treatment group. Patients in the control group will be given a home program by the orthopedic surgeon (common practice). Patients in the intervention (treatment) group will be treated with conventional physiotherapy 3 times a week for 6 weeks (4 times evaluation and 18 times treatment). all participants will be examined by the responsible examiner in physiotherapy clinic (blinded to the allocated group) at four main points: preoperative, postoperative (after the removal of spica cast), 3 weeks postoperative, 6 weeks postoperative.
Who Masked: Investigator, Outcomes Assessor
Masking Description: the primary investigator and the outcome assessor will assess all of the patients and will be blinded to the groups allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): this group will be treated as per the common practice postoperatively and will have the home program prescribed by the orthopedic surgeon
- intervention (treatment) group (Experimental): Patients in the intervention group will be treated with conventional physiotherapy 3 times a week for 6 weeks (18 times treatment).
  Interventions: Other: prescribed physiotherapy course

INTERVENTIONS:
Other: prescribed physiotherapy course — provide full assessment and treatment program as postoperative rehabilitation management
  Arms: intervention (treatment) group

SUMMARY:
Developmental Dysplasia of the Hip (DDH) is a common condition among young children that could range in severity. in most sever cases, surgical intervention is the best choice to correct the hip abnormality with the aim of restoring optimal functional ability. Referring patient for physiotherapy treatment post operative is not a common practice and surgeons relay on children natural developmental milestone in their recovery. however, prescribed physiotherapy treatment could promote maximum functional recovery and wellness. the aim of this research is (1) to evaluate the functional deference between patients who had conventional physiotherapy treatment program and patients who had home program prescribed by the orthopedic surgeon (2) to investigate what might be the underlying risk factors that could enhance or prohibit satisfactory functional level post operatively.

all individuals diagnosed with DDH and operated by Dr. Saleh Alsaifi (an orthopedic surgeon at alrazi orthopedic hospital) will be invited to participate in this study. The study will look at the children development in fictional ability postoperatively. not being referred to physiotherapy is a common practice, so the patients in the intervention group will benefit from having regular physiotherapy treatment with no risk at all. the study run from Alrazi orthopedic hospital in kuwait. the research is a collaboration between an orthopedic surgeon (Dr. Saleh Alsaifi) and physiotherapy team and it is expected to recruit all of the eligible patients through 12 months period (approximately 50 patients) then, the data will be sorted for analysis and reporting. the study is not funded with no personal interest.

DETAILED DESCRIPTION:
The population of the study: individuals diagnosed with DDH and operated by the orthopedic surgeon. Surgical procedures will include: open reduction, pelvic osteotomy (DEGA osteotomy) with/without femoral shortening. Individuals with operated DDH will be divided into two groups as conventional physiotherapy group and home program group. It will be ensured that the distribution of the individuals in the groups in a randomized manner, with the disease grades and operative procedures of the two treatment groups being the same and the clinical characteristics are similar.

The study will consist of children aged 1.5-5 who's guardian voluntarily agreed to participate in the study. It is planned to involve up to 50 children. Individuals who meet the inclusion criteria and had their guardian agreed to volunteer will be included in the study by signing the Informed Voluntary Consent Form. The participants will be examined by the responsible examiner in physiotherapy clinic (blinded to the allocated group). Patients in the control group will be given a home program by the orthopedic surgeon (common practice). Patients in the intervention group will be treated with conventional physiotherapy 3 times a week for 6 weeks (4 times evaluation and 18 times treatment).

As an outcome measure, the examiner will evaluate patient's hip function (using modified outcome evaluation standard for congenital dislocation of the hip by Zhou and Ji) and pediatric balance scale. patient will have a baseline data preoperatively. Then, patient will have the first postoperative evaluation10 weeks post-operatively (time of the removal of spica cast). After the first post-operative evaluation, individuals will be treated 3 times a week for 3 weeks and then the first evaluations will be done again then the same process will be repeated. Thus, Patient will be evaluated four times by the same examiner (before the operation, after 10 weeks [removal of spica cast], after 3 weeks of treatment [13 weeks postoperatively] and after 6 weeks of treatment [16 weeks postoperatively]). The data obtained before and after treatment and the data between the two groups will be compared.

Primary outcome measure modified outcome evaluation standard for congenital dislocation of the hip by Zhou will be used to evaluate child's functional level and Ji and pediatric balance scale will be used to evaluate child's balance. both outcome measures will be through physical examination of hip joint range of motion and some physical examination. the tests will be obtained 4 times (preoperative, postoperative base line (after the removal of the spica cast), 3 weeks post operative, 6 weeks postoperative)

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with DDH Tonnis grade 1-4 operated for open reduction, osteotomy with/without femoral shortening.
* patient is able to walk preoperatively
* aged between 1.5-5

Exclusion Criteria:

* Operated for DDH correction previously
* patient with neurological involvement
* patient with other congenital deformity
* patient with cognitive problems

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
modified outcome evaluation standard for congenital dislocation of the hip by Zhou and Ji will be used to evaluate child's functional level | Patient will be evaluated before the operation (baseline)
  evaluate the hip functional ability will start by measuring the hip range of motion in degrees and then graded from 0-5 where 5 is patient is able to do 100% of normal range of motion and 0 is less than 60% of normal ROM. this assessment will evaluate the hip flexion (normal ROM is 130-140),Hip abduction in extension position (normal ROM is 70),Hip abduction in flexion position (normal ROM is30-45), hip abduction (normal ROM is 20-30),Hip internal rotation (normal ROM is 40-50),Hip external rotation (normal ROM is 30-40). further more, the assessment tool will evaluate the pain ( in the scale of no, occasional, frequently), squat (normal, mildly, difficult), limping (none, mild, sever),Trendelenburg (negative, mild, positive), and shortening (none, mild<2cm, sever>2cm).
modified outcome evaluation standard for congenital dislocation of the hip by Zhou and Ji will be used to evaluate child's functional level | Patient will be evaluated after 10 weeks (removal of spica cast)
  evaluate the hip functional ability will start by measuring the hip range of motion in degrees and then graded from 0-5 where 5 is patient is able to do 100% of normal range of motion and 0 is less than 60% of normal ROM. this assessment will evaluate the hip flexion (normal ROM is 130-140),Hip abduction in extension position (normal ROM is 70),Hip abduction in flexion position (normal ROM is30-45), hip abduction (normal ROM is 20-30),Hip internal rotation (normal ROM is 40-50),Hip external rotation (normal ROM is 30-40). further more, the assessment tool will evaluate the pain ( in the scale of no, occasional, frequently), squat (normal, mildly, difficult), limping (none, mild, sever),Trendelenburg (negative, mild, positive), and shortening (none, mild<2cm, sever>2cm).
modified outcome evaluation standard for congenital dislocation of the hip by Zhou and Ji will be used to evaluate child's functional level | Patient will be evaluated after 3 weeks of treatment (13 weeks postoperatively)
  evaluate the hip functional ability will start by measuring the hip range of motion in degrees and then graded from 0-5 where 5 is patient is able to do 100% of normal range of motion and 0 is less than 60% of normal ROM. this assessment will evaluate the hip flexion (normal ROM is 130-140),Hip abduction in extension position (normal ROM is 70),Hip abduction in flexion position (normal ROM is30-45), hip abduction (normal ROM is 20-30),Hip internal rotation (normal ROM is 40-50),Hip external rotation (normal ROM is 30-40). further more, the assessment tool will evaluate the pain ( in the scale of no, occasional, frequently), squat (normal, mildly, difficult), limping (none, mild, sever),Trendelenburg (negative, mild, positive), and shortening (none, mild<2cm, sever>2cm).
modified outcome evaluation standard for congenital dislocation of the hip by Zhou and Ji will be used to evaluate child's functional level | Patient will be evaluated after 6 weeks of treatment (16 weeks postoperatively)
  evaluate the hip functional ability will start by measuring the hip range of motion in degrees and then graded from 0-5 where 5 is patient is able to do 100% of normal range of motion and 0 is less than 60% of normal ROM. this assessment will evaluate the hip flexion (normal ROM is 130-140),Hip abduction in extension position (normal ROM is 70),Hip abduction in flexion position (normal ROM is30-45), hip abduction (normal ROM is 20-30),Hip internal rotation (normal ROM is 40-50),Hip external rotation (normal ROM is 30-40). further more, the assessment tool will evaluate the pain ( in the scale of no, occasional, frequently), squat (normal, mildly, difficult), limping (none, mild, sever),Trendelenburg (negative, mild, positive), and shortening (none, mild<2cm, sever>2cm).
pediatric balance scale | Patient will be evaluated before the operation (baseline)
  the pediatric balance scale will evaluate the child's balance through asking the child to do 14 different tasks that include
  1. sitting to standing
  2. standing to sitting
  3. transfers.
  4. standing unsupported
  5. sitting unsupported
  6. standing with eyes closed
  7. standing with feet together.
  8. standing one foot in front
  9. standing on one foot
  10. turning 360 degrees
  11. turning to look behind
  12. retrieving object from the floor
  13. placing alternate foot on a stool
  14. reaching forward with outstretched arm. each task will be scored utilizing the 0-4 scale. the child's performance should be scored based upon the lowest criteria which describe the child best performance (each task has its own criteria of performance description scored from 0-4 that will be used to guide scoring procedure).
pediatric balance scale | Patient will be evaluated after 10 weeks (removal of spica cast)
  the pediatric balance scale will evaluate the child's balance through asking the child to do 14 different tasks that include
  1. sitting to standing
  2. standing to sitting
  3. transfers.
  4. standing unsupported
  5. sitting unsupported
  6. standing with eyes closed
  7. standing with feet together.
  8. standing one foot in front
  9. standing on one foot
  10. turning 360 degrees
  11. turning to look behind
  12. retrieving object from the floor
  13. placing alternate foot on a stool
  14. reaching forward with outstretched arm. each task will be scored utilizing the 0-4 scale. the child's performance should be scored based upon the lowest criteria which describe the child best performance (each task has its own criteria of performance description scored from 0-4 that will be used to guide scoring procedure).
pediatric balance scale | Patient will be evaluated after 3 weeks of treatment (13 weeks postoperatively)
  the pediatric balance scale will evaluate the child's balance through asking the child to do 14 different tasks that include
  1. sitting to standing
  2. standing to sitting
  3. transfers.
  4. standing unsupported
  5. sitting unsupported
  6. standing with eyes closed
  7. standing with feet together.
  8. standing one foot in front
  9. standing on one foot
  10. turning 360 degrees
  11. turning to look behind
  12. retrieving object from the floor
  13. placing alternate foot on a stool
  14. reaching forward with outstretched arm. each task will be scored utilizing the 0-4 scale. the child's performance should be scored based upon the lowest criteria which describe the child best performance (each task has its own criteria of performance description scored from 0-4 that will be used to guide scoring procedure).
pediatric balance scale | Patient will be evaluated after 6 weeks of treatment (16 weeks postoperatively)
  the pediatric balance scale will evaluate the child's balance through asking the child to do 14 different tasks that include
  1. sitting to standing
  2. standing to sitting
  3. transfers.
  4. standing unsupported
  5. sitting unsupported
  6. standing with eyes closed
  7. standing with feet together.
  8. standing one foot in front
  9. standing on one foot
  10. turning 360 degrees
  11. turning to look behind
  12. retrieving object from the floor
  13. placing alternate foot on a stool
  14. reaching forward with outstretched arm. each task will be scored utilizing the 0-4 scale. the child's performance should be scored based upon the lowest criteria which describe the child best performance (each task has its own criteria of performance description scored from 0-4 that will be used to guide scoring procedure).

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Hadeel Alsaleh, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: Yes
anonymous data will be shared for analysis
Supporting Information: SAP
Time Frame: Feb-April 2023 data will be destroyed after publication
Access Criteria: original data will be stored in a curly locked file section and only the primary investigator will have an access to this data.